CLINICAL TRIAL: NCT02715947
Title: Pharmacogenomics Study on Treatment of Psoriasis Vulgaris by Methotrexate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yijing He, Associate Professor, Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016 MTX/CSU/PS
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2015-12

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis Vulgaris; Methotrexate
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm (Experimental): intervention: open registry, non-randomized, single-arm trial.Methotrexate:2.5mg per piece, oral.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — During The first week: 7.5mg per week, oral; The second and third weeks: 10mg per week, oral; The fourth and fifth weeks: 12.5mg per week,oral; The sixth week:15mg per week, and maintain this dose, oral.
  Other Names: Amethopterin

SUMMARY:
To investigate the influence of genetic factors on the curative effect , to find the relationships between genetic variants and the response of Methotrexate to treatment of Psoriasis Vulgaris.

DETAILED DESCRIPTION:
Previous studies have indicated that the gene mutations of absorption distribution metabolism and drug target may affect the efficacy of Methotrexate in vivo.To investigate the influence of genetic factors on the curative effect , to find the relationships between genetic variants and the response of Methotrexate to treatment of Psoriasis Vulgaris.Investigators analyzed the various levels of genetic factors, including: 1.To analysis the key gene variants which associated with ADME(absorption, distribution, metabolism and excretion) affect the efficacy of Methotrexate; 2.Direct full genetic sequencing of MHC genes, to explore the genetic variations of efficacy and side effects; 3. Direct sequencing of all exons in the gene in the patients of the response of serious and effectively, to explores the rare genetic variation may cause deterioration of treatment by Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed according to Classification criteria for Psoriasis vulgaris
2. Patients aged 18 to 70 years (to the date of screening)
3. Not treatment in the Topical corticosteroids, Biologicals agents or Tretinoin cream
4. Phototherapy nearly one months before enrolled
5. Total bilirubin < 1.5 x ULN, AST(SGOT)/ALT(SGPT) <2.5 x ULN, if not liver metastases < 5 x ULN, if known liver metastases, Creatinine clearance <1.5 x ULN
6. Understanding the whole process of the study, voluntary participation and signed the informed consent

Exclusion Criteria:

1. Pregnant women, ready to pregnant or lactating women
2. Have a serious heart, lung, kidney and other vital organs and endocrine system lesions and the history
3. Patients is liver function abnormal persons (ALT above the center laboratory normal limit) or hepatitis b patient grain carriers
4. Patients with chronic diarrhea, or peptic ulcer nearly 1 year
5. Patients suffering from malignant tumor
6. Patients suffering from acute and chronic infectious diseases
7. Mental disorders, history of alcohol abuse, drug or other substance abuse
8. Other cases which researchers believe that can not enroll

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
disease control rate | 8 weeks after the first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, MD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided